CLINICAL TRIAL: NCT00990704
Title: Phase II, Open Study, Exploratory Examination of Efficacy and Safety of Paricalcitol Injection and Maxacalcitol Injection in Chronic Kidney Disease Subjects Receiving Hemodialysis With Secondary Hyperparathyroidism
Brief Title: Paricalcitol Compared to Maxacalcitol in Chronic Kidney Disease Patients With Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Yoshihiko Ueki, Abbott
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M11-609
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-06

CONDITIONS: Secondary Hyperparathyroidism; Hemodialysis
Keywords: Secondary hyperparathyroidism; Hemodialysis; paricalcitol; maxacalcitol
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — paricalcitol; maxacalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol (Experimental): 2 mcg adjusted by +/- 1 mcg, up to a maximum of 7 mcg, administered 3 times per week through intravenous catheter immediately before completion of dialysis
  Interventions: Drug: paricalcitol
- Maxacalcitol (Active Comparator): 5 or 10 mcg adjusted by +/- 2.5 mcg, up to a maximum of 20 mcg, administered 3 times per week through intravenous catheter immediately before completion of dialysis
  Interventions: Drug: maxacalcitol

INTERVENTIONS:
Drug: paricalcitol — Intravenous administration 3 times a week immediately before completion of dialysis
  Other Names: ABT-358; Zemplar
  Arms: Paricalcitol
Drug: maxacalcitol — Intravenous administration 3 times a week immediately before completion of dialysis
  Arms: Maxacalcitol

SUMMARY:
This study is a exploratory comparison of the efficacy and safety of paricalcitol injection with maxacalcitol injection in chronic kidney disease participants receiving hemodialysis with secondary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease (CKD) patients with iPTH >=300 pg/mL, adjusted calcium >=8.4 to <10.2 mg/dL, and phosphorus <=6.5 mg/dL
* Patients receiving dialysis 3 times weekly for at least 3 months before informed consent was obtained and scheduled to receive the same hemodialysis during the study period
* Patients using dialysate with constant concentration of calcium for 4 weeks before informed consent was obtained and receiving phosphate binder with constant dose regimen for 2 weeks before informed consent was obtained

Exclusion Criteria:

* Patients taking drugs that affect iPTH, calcium, or bone metabolism
* Patients with a history of allergic reaction or significant sensitivity to vitamin D
* Patients who received parathyroidectomy or ethanol infusion within 1 year before informed consent was obtained
* Patients with malignancy or with clinically significant hepatic disease (liver function tests more than 3 times the upper limit of normal) or with refractory hepatic disease
* Patients with cardiovascular disease designated as New York Heart Association Class III or IV or with any of the following cardiovascular or cerebrovascular diseases within 6 months before informed consent was obtained:

  * Acute coronary syndrome (myocardial infarction or unstable angina) or acute cerebral vascular disease (cerebral infarction or cerebral hemorrhage)
  * Coronary arterial revascularization (such as coronary artery bypass grafting, percutaneous transluminal coronary angioplasty)
  * Cerebral arterial revascularization (such as cerebral aneurysm clipping, cerebral aneurysm embolization, carotid artery endarterectomy)
  * Arteriosclerosis obliterans with rest pain (Fontaine classification III or more severe)
* Patients with severe hypertension (defined as mean resting blood pressure taken with the patient in a supine position before dialysis and at 6 dialyses sessions before informed consent was obtained: systolic >= 180 mmHg and diastolic >= 110 mmHg)
* Patients with uncontrolled diabetes mellitus (defined as mean glycosylated hemoglobin >=8% for 3 months before informed consent was obtained)
* Patients with a history of drug or alcohol abuse within 6 months before informed consent was obtained
* Patients who require chronic use of cytochrome P450 (CYP3A) inhibitors or inducers
* Patients who are taking products that contain aluminum 2 weeks before informed consent was obtained
* Patients who have taken paricalcitol in the past

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moriaki Kubo, Study Director — Abbott Japan Co.,Ltd
Locations (14):
- Japan (14):
  - Site Ref # / Investigator 53794, Anjo
  - Site Ref # / Investigator 53787, Chiba
  - Site Ref # / Investigator 53786, Kumagaya
  - Site Ref # / Investigator 53792, Matsumoto
  - Site Ref # / Investigator 53784, Mito
  - Site Ref # / Investigator 53796, Nagasaki
  - Site Ref # / Investigator 53795, Osaka
  - Site Ref # / Investigator 21561, Sapporo
  - Site Ref # / Investigator 53789, Tokyo
  - Site Ref # / Investigator 53790, Tokyo
  - Site Ref # / Investigator 53793, Toyohashi
  - Site Ref # / Investigator 53785, Tsuchiura
  - Site Ref # / Investigator 53788, Yachiyo
  - Site Ref # / Investigator 53791, Yokosuka

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Informed consent was obtained from 92 subjects; 45 of these subjects were not enrolled because they did not meet the eligibility criteria at the time of Screening.
Groups:
- Paricalcitol: 2 mcg with incremental of 1 mcg
- Maxacalcitol: 5 or 10 mcg with incremental of 2.5 mcg
Period: Overall Study
Arm/Group | Paricalcitol | Maxacalcitol
Started | 14 | 33
Completed | 13 | 31
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol | Maxacalcitol | Total
Number analyzed (Participants) | 14 | 33 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 19 | 25
  >=65 years | 8 | 14 | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 64.9 (11.02) | 61.5 (9.73) | 62.5 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 10 | 28 | 38
Region of Enrollment [Number; unit: participants]
  Japan | 14 | 33 | 47

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a >=50% Reduction in Intact Parathyroid Hormone (iPTH) From Baseline Compared to the Average iPTH Obtained in the Last 3 Weeks.
Time Frame: Baseline and the last 3 weeks (Weeks 11, 12, and 13)
Population: All subjects who received at least 1 dose of study drug and who had at least 1 iPTH measurement while on treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 14 | 33
Percentage of participants | 50.0 | 36.4
Statistical Analysis 1: Comparison: Paricalcitol vs Maxacalcitol; Test type: Superiority or Other; p = 0.518, Fisher Exact; Difference between arms in percentage = 13.6, 95% CI 2-sided [-22.36 to 49.63]

2. Secondary Outcome: The Percentage of Participants With iPTH Within Target Range of 60-180 pg/mL, Based on the Average iPTH Obtained in the Last 3 Weeks
Time Frame: During the last 3 weeks (Weeks 11, 12, and 13)
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 14 | 33
Percentage of participants | 28.6 | 15.2

3. Secondary Outcome: Mean iPTH at Each Visit
Time Frame: Screening (up to 2 weeks before Baseline) to Week 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 14 | 33
pg/mL
  Screening (up to 2 weeks before Baseline) | 462.7 (127.62) | 536.4 (190.72)
  Baseline (Week 1) | 507.6 (162.47) | 595.9 (213.80)
  Week 2 | 479.2 (178.43) | 474.8 (201.00)
  Week 3 | 474.4 (201.98) | 381.8 (181.07)
  Week 4 | 401.3 (209.24) | 310.2 (158.68)
  Week 5 | 373.2 (181.64) | 279.7 (155.07)
  Week 6 | 304.8 (136.76) | 262.3 (144.72)
  Week 7 | 282.2 (152.76) | 292.8 (187.02)
  Week 8 | 256.9 (142.39) | 315.1 (229.53)
  Week 9 | 275.9 (158.39) | 358.8 (252.98)
  Week 10 | 312.6 (140.45) | 361.2 (228.37)
  Week 11 | 279.6 (159.69) | 345.1 (189.52)
  Week 12 | 291.5 (163.51) | 341.6 (192.65)
  Week 13 | 293.0 (164.74) | 326.4 (180.33)

4. Secondary Outcome: Mean Change in iPTH From Baseline to the Average iPTH Obtained in the Last 3 Weeks
Time Frame: Baseline and the last 3 weeks (Weeks 11, 12, and 13)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 14 | 33
pg/mL | -208.4 (136.70) | -240.4 (152.73)

5. Secondary Outcome: Percentage of Participants With a >= 50% Reduction in iPTH From Baseline to the Average iPTH Obtained in the Last 3 Weeks and Without Hypercalcemia During Treatment
Description: Hypercalcemia was defined as at least 1 corrected calcium > 11.5 mg/dL or at least 2 consecutive corrected calcium >= 11.0 mg/dL.
Time Frame: Baseline and the last 3 weeks (Weeks 11, 12, and 13) for iPTH and anytime during the 12-week treatment period for hypercalcemia
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 14 | 33
Percentage of participants | 50.0 | 33.3

6. Secondary Outcome: Percentage of Participants With iPTH Within the Target Range of 60-180 pg/mL Based on the Average iPTH Obtained in the Last 3 Weeks of the Study and Without Hypercalcemia Anytime During Treatment
Description: as for outcome 5
Time Frame: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 14 | 33
Percentage of participants | 28.6 | 12.1

7. Secondary Outcome: Number of Occurrences of iPTH Control, Defined as >=50% Reduction in iPTH From Baseline
Time Frame: Over the 12-week treatment period
Measure: Mean (Standard Deviation); unit: Occurrences per participant
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 14 | 33
Occurrences per participant | 3.4 (2.98) | 4.8 (2.96)

8. Secondary Outcome: Number of Occurrences of iPTH Control, Defined as Within the Target Range of 60-180 pg/mL of iPTH
Time Frame: Over the 12-week treatment period
Measure: Mean (Standard Deviation); unit: Occurrences per participant
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 14 | 33
Occurrences per participant | 2.3 (2.70) | 2.7 (2.67)

ADVERSE EVENTS:
Arm/Group | Paricalcitol | Maxacalcitol
Serious Adverse Events (participants affected / at risk) | 3/14 | 3/33
Other Adverse Events (participants affected / at risk) | 14/14 | 31/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=14) | Maxacalcitol (N=33)
Cataract (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Pyothorax (Injury, poisoning and procedural complications) | 1 | 0
Skin papilloma (Skin and subcutaneous tissue disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=14) | Maxacalcitol (N=33)
Eye pruritus (Eye disorders) | 1 | 0
Scleritis (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 1 | 1
Gingivitis (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Stomach discomfort (Gastrointestinal disorders) | 0 | 2
Injection site dermatitis (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 12
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 2 | 4
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 1
Blood pressure decreased (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Skin chapped (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 2
Hypertension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.